CLINICAL TRIAL: NCT04364997
Title: A Multi-center, Randomized, Double-blind, Double-simulation, Duloxetine Hydrochloride Enteric-coated Positive-control Phase III Study of Desvenlafaxine Succinate Sustained-Release in the Treatment of Major Depressive Disorder.
Brief Title: Study of Desvenlafaxine in Treating Major Depressive Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HF124-CSP-001
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Desvenlafaxine
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desvenlafaxine Succinate Sustained-Release (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release Tablet , Duloxetine Hydrochloride Enteric-coated Capsule Placebo; Drug: Duloxetine Hydrochloride Enteric-coated Capsule Placebo
- Duloxetine Hydrochloride Enteric-coated (Active Comparator)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release Tablet Placebo, Duloxetine Hydrochloride Enteric-coated Capsule; Drug: Duloxetine Hydrochloride Enteric-coated Capsule

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release Tablet , Duloxetine Hydrochloride Enteric-coated Capsule Placebo — Desvenlafaxine Succinate Sustained-Release Tablet 50 mg+Duloxetine Hydrochloride Enteric-coated Capsule Placebo 60 mg orally once daily for 8 weeks.
  Arms: Desvenlafaxine Succinate Sustained-Release
Drug: Desvenlafaxine Succinate Sustained-Release Tablet Placebo, Duloxetine Hydrochloride Enteric-coated Capsule — Desvenlafaxine Succinate Sustained-Release Tablet Placebo 50mg +Duloxetine Hydrochloride Enteric-coated Capsule 60mg orally once daily for 8 weeks,
  Arms: Duloxetine Hydrochloride Enteric-coated
Drug: Duloxetine Hydrochloride Enteric-coated Capsule Placebo — Duloxetine Hydrochloride Enteric-coated Capsule Placebo 30 mg orally once daily for 1 week after 8-weeks treatment.
  Arms: Desvenlafaxine Succinate Sustained-Release
Drug: Duloxetine Hydrochloride Enteric-coated Capsule — Duloxetine Hydrochloride Enteric-coated Capsule 30mg orally once daily for 1 week after 8-weeks treatment.
  Arms: Duloxetine Hydrochloride Enteric-coated

SUMMARY:
The primary purpose of this study is to evaluate if the effectiveness of desvenlafaxine succinate sustained-release tablet (50 mg/day) used for 8 weeks is not inferior to duloxetine hydrochloride enteric-coated capsule (60 mg/day) in adult patients with major depressive disorder.

DETAILED DESCRIPTION:
This is a multicenter study to evaluate if the effectiveness of desvenlafaxine succinate sustained-release tablet (50 mg/day) used for 8 weeks is not inferior to duloxetine hydrochloride enteric-coated capsule (60 mg/day) in adult patients with major depressive disorder. A total of 400 subjects will be randomly allocated to experimental arm (desvenlafaxine succinate sustained-release tablet) and active comparator arm (duloxetine hydrochloride enteric-coated capsule) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 65 years old, male or female;
* Outpatients and inpatients who met the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria and Neuropsychiatric Interview5.0.0 (MINI5.0.0) for a primary diagnosis of Major Depressive Disorder(MDD), single or recurrent episode and measured by the Mini-International Neuropsychiatric Interview5.0.0 (MINI5.0.0) as active stage.
* Hamilton Psychiatric Rating Scale for Depression (HAM-D17) total score of >= 18.

Exclusion Criteria:

* Hamilton Rating Scale for Anxiety (HAM-A) total score of > 14.
* Refractory depression: Ineffective after adequate treatment with two or more antidepressants.
* Current or previous diagnosis of Axis I with DSM-IV other than depression.
* Significant risk of suicide based on clinical judgment or HAM-D 17, Suicide attempt in the past 6 months.
* Any unstable hepatic, renal, pulmonary, cardiovascular (including uncontrolled hypertension), ophthalmologic, neurologic, or any other medical condition that might confound the study or put the subject at greater risk during study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Change From Baseline on the Hamilton Rating Scale for Depression, 17-item Total Score (HAM-D17) at Week 8 | Baseline to Week 8
  Hamilton Rating Scale for Depression, 17-item is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Each item is scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), for a maximum total score of 52; higher scores indicate more depression. Change from baseline: score at observation minus score at baseline.

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression, 17-item (HAM-D17) Response Rate | Baseline to Week 8
  Hamilton Rating Scale for Depression, 17-item is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Each item is scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), for a maximum total score of 52; higher scores indicate more depression. A response is defined as ≥ 50% decrease from baseline on Hamilton Psychiatric Rating Scale for Depression (HAM-D17) total score.
Hamilton Rating Scale for Depression, 17-item (HAM-D17) Remission Rate | Baseline to Week 8
  Hamilton Rating Scale for Depression, 17-item is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Each item is scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), for a maximum total score of 52; higher scores indicate more depression. Remission is defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) total score of ≤ 7.
Change From Baseline on the Hamilton Rating Scale for Anxiety (HAM-A) Total Score | Baseline to Week 8
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale which consists of 14 items, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The highest possible score is 56, which represents the most severe form of anxiety; the lowest possible score is 0, which represents an absence of anxiety.
Change From Baseline on the Clinical Global Impression Scale-Improvement (CGI-I) | Baseline to Week 8
  Clinical Global Impression Scale-Improvement (CGI-I): 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Higher score = worse outcome.
Change From Baseline on the Clinical Global Impression-Severity Score (CGI-S) | Baseline to Week 8
  Clinical Global Impression-Severity Score (CGI-S): 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = worse state.
Change From Baseline on the Visual Analog Scale (VAS) for Pain | Baseline to Week 8
  The pain level was assessed with the Visual Analog Scale, which consists of a horizontal line of 10 cm in length. For pain level assessment, "0" defines "no pain" and "10" defines "unbearable pain''. The participants are asked to mark the intensity of their pain level.

CONTACTS AND LOCATIONS:
Overall Officials: Xuefang Xia, Study Chair — Department of Medicine, CSPC Clinical Development Division
Locations (1):
- Beijing Anding Hospital, Beijing, China